CLINICAL TRIAL: NCT00643929
Title: LENS - Long-term Eltrombopag Observational Study - A Long Term Observational Ocular Safety Follow-up Study in Adults Who Have Received Study Medication (SB-497115-GR / Eltrombopag Olamine or Placebo) in a Phase II or III Clinical Study Evaluating Eltrombopag
Brief Title: LENS - Long-term Eltrombopag Observational Study
Acronym: LENS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: TRA108132
Record Dates: First submitted 2008-03-06; First posted 2008-03-26 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: thrombopoietin receptor agonist; ocular safety; HCV; SB-497115-GR; CIT; ITP; cataract; eltrombopag olamine; lens opacity
MeSH Terms: conditions — Purpura; Cataract | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Subjects who have participated in a prior eltrombopag study, receiving either placebo or eltrombopag
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Subjects participated in a prior eltrombopag study, having received either eltrombopag or placebo
  Other Names: Promacta

SUMMARY:
A long term observational ocular safety study in adults who have received study medication (either active drug or placebo) in a phase II or III clinical study evaluating eltrombopag. The study will follow subjects for 2.5 years following their last ocular assessment on their prior treatment study (regardless of the therapeutic indication) and will describe long-term ocular safety with respect to changes in the lenses over time from all subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for enrolment in the study if they have previously participated in an eltrombopag study, either phase II or III, and meet all of the following criteria:

* Subject has signed and dated a written informed consent for this study.
* Subject has previously participated in a study evaluating eltrombopag, either phase II or III, and must have received at least one dose of study medication (either active drug or placebo). This excludes subjects from phase I studies (See Section 5.1).
* The prescribed follow-up ophthalmic assessment at 6 months post end of treatment should be completed as specified in the protocol for the previous study.
* Subject is able to understand and comply with protocol requirements and instructions.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Subject has received surgery for cataracts and is aphakic or bilaterally pseudophakic.
* In some countries (i.e. France), a subject is neither affiliated with nor a beneficiary of a social security category.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who participated in a prior eltrombopag study, regardless of indication, and have received either placebo or eltrombopag.
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2007-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Description of the incidence of changes in lens over time | 2.5 years

SECONDARY OUTCOMES:
Exploratory epidemiologic analyses of ocular data from patients previously enrolled in studies with eltrombopag. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (63):
- United States (5):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Richmond, Virginia
- GSK Investigational Site, Kogarah, New South Wales, Australia
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Canada (5):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Montreal, Quebec
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
- France (7):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- GSK Investigational Site, Berlin, State of Berlin, Germany
- GSK Investigational Site, Shatin, New Territories, Hong Kong
- GSK Investigational Site, Budapest, Hungary
- India (4):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mumbai
- Italy (6):
  - GSK Investigational Site, San Giovanni Rotondo, Apulia
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
- GSK Investigational Site, Karachi, Pakistan
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Lima
- GSK Investigational Site, Poznan, Poland
- GSK Investigational Site, San Juan, Puerto Rico, Puerto Rico
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, St'Petersburg
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- GSK Investigational Site, Stockholm, Sweden
- Tunisia (4):
  - GSK Investigational Site, Montfleury
  - GSK Investigational Site, Sfax
  - GSK Investigational Site, Sousse
  - GSK Investigational Site, Tunis
- Ukraine (4):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Vinnytsia
- United Kingdom (4):
  - GSK Investigational Site, Plymouth, Devon
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, London
  - GSK Investigational Site, Morriston